CLINICAL TRIAL: NCT05522842
Title: Evaluation of Corneal Endothelium in Diabetic Patients Undergoing Phacoemulsification Using Specular Microscopy
Brief Title: Corneal Endothelium in Diabetics Undergoing Phacoemulsification
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rahma Rashad Helmy, doctor, Assiut University
Other Study IDs: corneal endothelium
Record Dates: First submitted 2022-08-13; First posted 2022-08-31 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-09

CONDITIONS: Corneal Endothelial Cell Loss
MeSH Terms: conditions — Corneal Endothelial Cell Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
evaluate and compare the changes in corneal endothelial cell count density between diabetic and non diabetic patients undergoing phacoemulsification surgery, and to evaluate the effect of duration, and control of diabetes on corneal morphology.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a major health hazard reaching epidemic proportions. Worldwide more than 285 million people are affected by DM; this number is expected to increase to 439 million by 2030 according to the international diabetes federation. DM affects every part of the body and the eye is not an exception.

Diabetes mellitus has been found to be detrimental to corneal endothelium . Patients with diabetes have been found to have morphologically abnormal endothelium, including pleomorphism and polymegethism. Also, elderly patients with diabetes mellitus undergo phacoemulsification is particularly vulnerable to greater endothelial damage during surgery than non diabetics.

Several studies showed that diabetes mellitus has a lower impact on corneal cell density and morphology in patients with good glycemic control , also patients with diabetes over 10 years have more corneal morphological abnormalities than those having diabetes under 10 years duration.

Patients with DM tend to develop cataract more frequently and earlier than non diabetics.

Corneal endothelium plays an important role in maintaining dehydrated state and transparency of cornea throughout life, by pumping excess fluid out of stroma through active transport mechanism and barrier function. Any compromise in these factors leads to direct effect on corneal endothelium .

Cataract has been documented to be the most significant cause of bilateral blindness .

Cataract extraction with phacoemulsification is one of the most common surgical procedure performed nowadays, with an estimated 19 million operation performed annually worldwide. The WHO states that this number will increase to 32 million by 2025, however corneal endothelium is known to undergo damage during phacoemulsification in many different ways, it may be injured mechanically as result of instrumentation causing postoperative complication such as corneal edema.

Specular microscopy is used for non invasive viewing and recording of the image of corneal endothelial cell layer. Several studies have used specular microscopy for quantitative assessment of the corneal damage associated with phacoemulsification by measuring the degree of decrease in the corneal cell density.

ELIGIBILITY:
Inclusion Criteria:

* Age from 40 to 70
* Any degree of cataract
* No previous ocular surgery

Exclusion Criteria:

* Any corneal pathology, infection, or active inflammation
* pseudoexofoliation
* History of ocular trauma or surgery

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: evaluate the changes in corneal endothelium between 50 patients diabetic and non diabetic undergoing phacoemulsification
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
corneal endothelium cell count | baseline
  normal range of 1500 to 3500 cells/mm2 (age, 40-90)
corneal endothelial cell size | baseline
  their dimension being roughly 50-70 μm long, 10-30 μm wide and 0.1-10 μm thick
corneal endothelial cell shape | baseline
  a single layer of cells organized in a characteristic honeycomb pattern